CLINICAL TRIAL: NCT02142868
Title: AN EXPANDED ACCESS STUDY OF PALBOCICLIB IN COMBINATION WITH LETROZOLE AS TREATMENT OF POST-MENOPAUSAL WOMEN WITH HORMONE RECEPTOR POSITIVE, HER2 NEGATIVE ADVANCED BREAST CANCER FOR WHOM LETROZOLE THERAPY IS DEEMED APPROPRIATE
Brief Title: Expanded Access Study Of Palbociclib (PD-0332991) In Combination With Letrozole As Treatment Of Post-Menopausal Women With HR-Positive, Her2-Negative Advanced Breast Cancer For Whom Letrozole Therapy Is Deemed Appropriate
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481034
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Advanced Breast Cancer (Female)
Keywords: Expanded Access; Advanced Breast Cancer
MeSH Terms: interventions — palbociclib; Letrozole

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered orally once a day at 125 mg/day for 21 days followed by 7 days off treatment for each 28-day cycle (Schedule 3/1)
  Other Names: Ibrance
Drug: Letrozole — Letrozole will be administered orally at 2.5 mg once daily as continuous daily dosing schedule according to product labeling and in compliance with its local prescribing information.
  Other Names: Femara

SUMMARY:
To provide access to palbociclib to post-menopausal women with HR-positive, HER2-negative advanced breast cancer who are deemed appropriate for letrozole therapy (Canada: first-line patients only).

DETAILED DESCRIPTION:
This study is currently available in Canada only.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women 18 years of age or above with proven diagnosis of advanced adenocarcinoma of the breast (locoregionally recurrent or metastatic disease)
* ER-positive and/or PR-positive tumor based on local laboratory results
* HER2-negative tumor based on local laboratory results
* Patients must be appropriate candidates for letrozole therapy (Canada: first-line patients only)

Exclusion Criteria:

* Patients who have previously participated in a palbociclib trial or who have received prior treatment with any CDK inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (40):
  - CBCC Global Research, Inc. at Comprehensive Blood & Cancer Center Research Center, Bakersfield, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Gwinnett Hospital System Inc. -d/b/a - The Center for Cancer Care, Duluth, Georgia
  - Gwinnett Hospital System Inc. -d/b/a - The Center for Cancer Care, Lawrenceville, Georgia
  - Presence Saint Joseph Hospital, Chicago, Illinois
  - North Shore Oncology-Hematology Associates, Ltd., Crystal Lake, Illinois
  - North Shore Oncology-Hematology Associates, Ltd., Libertyville, Illinois
  - Presence Medical Group Hematology Oncology, Northbrook, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Presence Infusion Care - Skokie, Skokie, Illinois
  - Metairie Oncologist, LLC, Metairie, Louisiana
  - SKCCC at Johns Hopkins, The Harry and Jeannette Weinberg Building, Baltimore, Maryland
  - SKCCC at Johns Hopkins, Green Spring Station, Lutherville, Maryland
  - The West Clinic, P.C., Corinth, Mississippi
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Mississippi Baptist Health Systems, Jackson, Mississippi
  - The West Clinic, P.C. d/b/a West Cancer Center, Southaven, Mississippi
  - ProHealthCARE Associates, LLP, Lake Success, New York
  - Northwest Cancer Specialists dba Compass Oncology, Portland, Oregon
  - UPMC Cancer Center Beaver, Beaver, Pennsylvania
  - UPMC Cancer Center Arnold Palmer at Mountainview, Greensburg, Pennsylvania
  - UPMC Cancer Center Greenville, Greenville, Pennsylvania
  - UPMC Cancer Center Monroeville, Monroeville, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Cancer Center St. Margarets, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Investigational Drug Service, William M. Cooper Pavilion, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, William M. Cooper Pavilion, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center Passavant (HOA), Pittsburgh, Pennsylvania
  - UPMC Cancer Center Passavant (OHA), Pittsburgh, Pennsylvania
  - UPMC Cancer Center Northwest, Seneca, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - The West Clinic, P.C. d/b/a West Cancer Center, Germantown, Tennessee
  - The West Clinic, P.C. d/b/a West Cancer Center, Memphis, Tennessee
  - Texas Oncology -Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Medical Oncology & Hematology Associates of Northern Virginia, Ltd., Fairfax, Virginia
  - Medical Oncology & Hematology Associates of Northern Virginia, Ltd., Reston, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Northwest Cancer Specialists dba Compass Oncology, Vancouver, Washington
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Holy Cross Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Queen Elizabeth II (QEII) Health Sciences Centre, Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook health Sciences Centre, Toronto, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - SunnyBrook Research Institute, Toronto, Ontario
  - McGill University Health Centre (MUHC), Glen Site, Royal Victoria Hospital, Cedars Cancer Centre, Montreal, Quebec
  - CHU de Quebec - Hospital du Saint-Sacrement, Québec, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/